CLINICAL TRIAL: NCT04162470
Title: An Open-label Extension Study to Evaluate the Long-term Safety, Tolerability, and Efficacy of REGN3918 in Patients With Paroxysmal Nocturnal Hemoglobinuria
Brief Title: REGN3918 in Patients With Paroxysmal Nocturnal Hemoglobinuria (PNH) to Evaluate Its Long Term Safety, Efficacy and Tolerability.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business Decision
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R3918-PNH-1868; 2019-000130-20 (EudraCT Number)
Record Dates: First submitted 2019-11-11; First posted 2019-11-14 (Actual); Results first posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-05

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
Keywords: PNH
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- REGN3918 (Experimental): Participants who have completed 1 of the 2 parent studies (R3918-PNH-1852 [NCT03946748] or R3918-PNH-1853)
  Interventions: Drug: REGN3918

INTERVENTIONS:
Drug: REGN3918 — Subcutaneous (SC) every week (QW) over the treatment period
  Other Names: Pozelimab

SUMMARY:
The primary objective of the study is to evaluate the long-term safety, tolerability, and effect on intravascular hemolysis of REGN3918 in patients with paroxysmal nocturnal hemoglobinuria (PNH).

The secondary objectives of the study are:

* To evaluate the long-term effect of REGN3918 on intravascular hemolysis
* To assess the concentrations of total REGN3918 in serum
* To evaluate the occurrence of the immunogenicity of REGN3918

ELIGIBILITY:
Key Inclusion Criteria:

• Patients with PNH who have completed, without discontinuation, study treatment in one of the parent studies in which they participated (either R3918-PNH-1852 [NCT03946748] or R3918-PNH-1853)

Key Exclusion Criteria:

* Significant protocol deviation(s) in the parent study based on the investigator's judgment and to the extent that these would (if continued) impact the study objectives and/or safety of the patient (for example, repetitive non-compliance with dosing by the patient)
* Any new condition or worsening of an existing condition which, in the opinion of the investigator, would make the patient unsuitable for enrollment or could interfere with the patient participating in or completing the study

NOTE: Other protocol defined exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2022-04-07 (Actual); Study Completion 2022-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (10):
- Regeneron Study Site, Shatin, Hong Kong
- Regeneron Study Site, Budapest, Hungary
- Malaysia (3):
  - Regeneron Study Site, Miri, Sarawak
  - Regeneron Study Site, Sibu, Sarawak
  - Regeneron Study Site, Kuala Terengganu, Terengganu
- South Korea (2):
  - Regeneron Study Site, Busan
  - Regeneron Study Site, Seoul
- Taiwan (2):
  - Regeneron Study Site, Taipei
  - Regeneron Study Site, Taoyuan
- Regeneron Study Site, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Individual anonymized participant data will be considered for sharing once the indication has been approved by a regulatory body, if there is legal authority to share the data and there is not a reasonable likelihood of participant re-identification.
Access Criteria: Qualified researchers may request access to anonymized patient level data or aggregate study data when Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency [EMA], Pharmaceuticals and Medical Devices Agency [PMDA], etc) for the product and indication, has the legal authority to share the data, and has made the study results publicly available (eg, scientific publication, scientific conference, clinical trial registry).
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the study, the sponsor made an administrative decision to terminate the pozelimab monotherapy program, all participants were withdrawn from this study.
Groups:
- REGN3918: Participants who completed parent study R3918-PNH-1852 (NCT03946748) received pozelimab 800 milligrams (mg) subcutaneous (SC) injection once weekly (QW) for up to 104 weeks.
Period: Overall Study
Arm/Group | REGN3918
Started | 24
Completed | 0
Not Completed | 24
Not completed — Withdrawn due to sponsor's decision | 24

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAF) included all enrolled participants who received any study drug.
Groups:
- REGN3918: Participants who completed parent study R3918-PNH-1852 (NCT03946748) received pozelimab 800 mg SC injection QW for up to 104 weeks.
Arm/Group | REGN3918
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.8 (17.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 21
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. TEAEs was defined as AEs that developed or worsened during the on-treatment period. SAE was defined as any untoward medical occurrence that resulted in any of following outcomes: death, life-threatening, required initial/prolonged in-participant hospitalization, persistent/significant disability/incapacity, congenital anomaly/birth defect/considered as medically important event. TEAEs included both Serious TEAEs and non-serious TEAEs.
Time Frame: Baseline up to Week 104
Population: SAF included all enrolled participants who received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | REGN3918
Number analyzed (Participants) | 24
Participants
  Participants with TEAEs | 15
  Participants with Serious TEAEs | 2

2. Primary Outcome: Percentage of Participants Who Achieved Lactate Dehydrogenase (LDH) Less Than or Equal to (≤) 1.5* ULN From Baseline to Week 26
Description: Percentage of participants who achieved LDH ≤1.5* Upper limit of normal (ULN) over Week 26, defined as LDH ≤1.5*ULN from baseline up to Week 26 were reported. A participant was considered to have met the criteria for adequate control of intravascular hemolysis if all of their LDH readings from the baseline through Week 26 inclusive or through the analysis end date, whichever is earlier, had values ≤ 1.5*ULN.
Time Frame: Baseline up to Week 26
Population: Full Analysis Set (FAS) included all enrolled participants who received any study drug. Here, "Overall number of Participants Analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | REGN3918
Number analyzed (Participants) | 23
Percentage of participants | 95.7 [87.3 to 100.0]

3. Secondary Outcome: Percentage of Participants Who Had Breakthrough Hemolysis Through Week 26 and 78
Description: A participant was considered to have breakthrough hemolysis if he/she had any LDH measurement greater than or equal to (≥) 2*ULN, concomitant with associated signs or symptoms at any time subsequent to an initial achievement of disease control (i.e., LDH ≤ 1.5* ULN).
Time Frame: At Week 26 and 78
Population: FAS included all enrolled participants who received any study drug. Here, "Overall number of Participants Analyzed" signifies participants who were evaluable for this outcome measure and "number analyzed" signifies those participants who were evaluable at the specified time points.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | REGN3918
Number analyzed (Participants) | 23
Percentage of participants
  At Week 26 | 0 [0 to 0]
  At Week 78: number analyzed (Participants) | 15
  At Week 78 | 0 [0 to 0]

4. Secondary Outcome: Overall Rate of Transfusion With Red Blood Cell (RBCs) Through Week 26
Description: The overall rate of transfusion for a participant was calculated based on the duration of treatment exposure of the participant.
Time Frame: Baseline up to Week 26
Population: FAS included all enrolled participants who received any study drug.
Measure: Number (95% Confidence Interval); unit: Transfusion per person-year of treatment
Arm/Group | REGN3918
Number analyzed (Participants) | 24
Transfusion per person-year of treatment | 0.164 [0.006 to 4.678]

5. Secondary Outcome: Percentage of Participants Who Are Transfusion-free (With RBCs) Through Week 26 and 78
Description: Transfusion free was defined as not having received an RBC transfusion during the first 26 and 78 weeks. A transfusion was counted only if it was per-protocol, that is, if it follows the predefined transfusion algorithm: RBC transfusion due to a post-baseline hemoglobin level less than (<) 9 gram per deciliter (g/dL) (with anemia symptoms) or a post-baseline hemoglobin level < 7 g/dL (without anemia symptoms).
Time Frame: At Week 26 and 78
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | REGN3918
Number analyzed (Participants) | 23
Percentage of participants
  At Week 26 | 95.7 [87.3 to 100.0]
  At Week 78: number analyzed (Participants) | 16
  At Week 78 | 93.8 [81.9 to 100.0]

6. Secondary Outcome: Percentage of Participants Who Achieved Adequate Control of Intravascular Hemolysis Through Week 78
Description: A participant was considered to have met the criteria for adequate control of intravascular hemolysis if all of his/her LDH readings from the baseline through Week 78 inclusive or through the analysis end date, whichever is earlier, had values <=1.5* ULN. and must not have discontinued study treatment early.
Time Frame: Baseline up to Week 78
Population: FAS included all enrolled participants who received any study drug. Here, "Overall number of Participants Analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | REGN3918
Number analyzed (Participants) | 16
Percentage of participants | 93.8 [81.9 to 100.0]

7. Secondary Outcome: Percentage of Participants Who Achieved Normalization of Intravascular Hemolysis Through Week 26 and Week 78
Description: A participant was considered to have met normalization of intravascular hemolysis if all of their LDH readings from the baseline through Week 26 or 78 inclusive, or through the analysis end date, whichever is earlier, had values ≤ 1.0*ULN.
Time Frame: Baseline, Week 26 and 78
Population: FAS included all enrolled participants who received any study drug. Here, "number analyzed" signifies those participants who were evaluable at the specified time points.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | REGN3918
Number analyzed (Participants) | 24
Percentage of participants
  At Week 26 | 75.0 [57.7 to 92.3]
  At Week 78: number analyzed (Participants) | 20
  At Week 78 | 55.0 [33.2 to 76.8]

8. Secondary Outcome: Changes From Baseline in LDH Levels at Week 26, 78, and 104
Description: Change from baseline in LDH levels at Week 26, 78, and 104 was reported. Reported baseline is from R3918-PNH-1852 study.
Time Frame: Baseline, Week 26, 78, and 104
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units per liter (U/L)
Arm/Group | REGN3918
Number analyzed (Participants) | 24
Units per liter (U/L)
  At Week 26 | -5.098 (2.5695)
  At Week 78: number analyzed (Participants) | 17
  At Week 78 | -5.395 (2.8468)
  At Week 104: number analyzed (Participants) | 15
  At Week 104 | -5.270 (2.9057)

9. Secondary Outcome: Percent Change From Baseline in LDH Levels at Week 26, 78, and 104
Description: Percent change from baseline in LDH levels at Week 26, 78, and 104 was reported. Reported baseline is from R3918-PNH-1852 study.
Time Frame: Baseline, Week 26, 78, and 104
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | REGN3918
Number analyzed (Participants) | 24
Percent change
  At Week 26 | -81.900 (8.9226)
  At Week 78: number analyzed (Participants) | 17
  At Week 78 | -84.256 (8.1412)
  At Week 104: number analyzed (Participants) | 15
  At Week 104 | -83.930 (7.6705)

10. Secondary Outcome: Change From Baseline in Red Blood Cell (RBC) Hemoglobin Levels at Week 26, 78, and 104
Description: Change from baseline in RBC hemoglobin levels at Week 26, 78, and 104 was reported.
Time Frame: Baseline, Week 26, 78, and 104
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Gram per liter (g/l)
Arm/Group | REGN3918
Number analyzed (Participants) | 21
Gram per liter (g/l)
  At Week 26 | 3.6 (8.97)
  At Week 78: number analyzed (Participants) | 14
  At Week 78 | 5.3 (17.20)
  At Week 104: number analyzed (Participants) | 5
  At Week 104 | -2.4 (16.56)

11. Secondary Outcome: Change From Baseline in Free Hemoglobin Levels at Week 26, 78 and 104
Description: Change from baseline in free hemoglobin levels at Week 26, 78 and 104 was reported.
Time Frame: Baseline, Week 26, 78 and 104
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Milligram per deciliter (mg/dL)
Arm/Group | REGN3918
Number analyzed (Participants) | 16
Milligram per deciliter (mg/dL)
  At Week 26 | -1.39 (6.929)
  At Week 78: number analyzed (Participants) | 7
  At Week 78 | -0.56 (2.196)
  At Week 104: number analyzed (Participants) | 4
  At Week 104 | -0.93 (1.153)

12. Secondary Outcome: Serum Concentrations of Total REGN3918
Description: Serum Concentrations of total REGN3918 was reported.
Time Frame: Pre-dose (Day 1), End of infusion at Week 13, 26, 39, 52, 65, 78, 91 and 104
Population: Here, "Overall number of Participants Analyzed" signifies participants who were evaluable for this outcome measure and "number analyzed" signifies those participants who were evaluable at the specified time points.
Measure: Mean (Standard Deviation); unit: Milligrams per liter (mg/L)
Arm/Group | REGN3918
Number analyzed (Participants) | 23
Milligrams per liter (mg/L)
  Pre-dose (Day 1) | 423 (218)
  Week 13 | 398 (203)
  Week 26 | 401 (212)
  Week 39: number analyzed (Participants) | 18
  Week 39 | 420 (216)
  Week 52: number analyzed (Participants) | 17
  Week 52 | 413 (202)
  Week 65: number analyzed (Participants) | 16
  Week 65 | 438 (207)
  Week 78: number analyzed (Participants) | 10
  Week 78 | 433 (266)
  Week 91: number analyzed (Participants) | 8
  Week 91 | 483 (278)
  Week 104: number analyzed (Participants) | 0

13. Secondary Outcome: Number of Participants With Treatment-emergent Anti-Drug Antibodies (ADA) to REGN3918
Description: Number of Participants with treatment-emergent ADA response to REGN3918 was reported.
  The ADA analysis set (AAS) includes all treated participants who received any amount of study drug (active [SAF]) and had at least 1 non missing anti pozelimab antibody result following the first dose of study drug. The AAS is based on the actual treatment received (as treated).
Time Frame: Baseline up to Week 104
Population: Here, "number analyzed" signifies those participants who were evaluable at the specified time points.
Measure: Count of Participants; unit: Participants
Arm/Group | REGN3918
Number analyzed (Participants) | 21
Participants | 0

ADVERSE EVENTS:
Time Frame: From first dose to Week 104
Arm/Group | REGN3918
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 2/24
Other Adverse Events (participants affected / at risk) | 6/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | REGN3918 (N=24)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | REGN3918 (N=24)
Mouth ulceration (Gastrointestinal disorders) | 2 (2)
Chills (General disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2019-03-19): https://cdn.clinicaltrials.gov/large-docs/70/NCT04162470/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-07): https://cdn.clinicaltrials.gov/large-docs/70/NCT04162470/SAP_001.pdf